CLINICAL TRIAL: NCT05900869
Title: Reduction Nymphoplasty: Assessment of the Impact on Sexuality, Self-Esteem and Screening for Dysmorphophobia
Acronym: NYRESED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NYRESED-Local/2023/JS-01
Record Dates: First submitted 2023-05-30; First posted 2023-06-13 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Plastic Surgery
MeSH Terms: interventions — BES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FSFI — Female Sexual Function Index questionnaire
Other: BES — Body Esteem Scale questionnaire

SUMMARY:
Reduction nymphoplasty is the treatment of benign hyperplasia of the labia minora. This surgery is indicated in the event of functional, aesthetic or sexual discomfort. There has been a growing demand for this surgery over the past twenty years. It is necessary to remain vigilant because a request for cosmetic surgery can also be part of an obsession with body dysmorphism, former dysmorphophobia.

Investigators wish to study the postoperative results concerning sexuality, self-esteem and obsession with body dysmorphia in a cohort of patients followed prospectively and at more than 3 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patients informed of the objectives of the study and its progress,

Exclusion Criteria:

Patients in a period of exclusion determined by another study. Patients under judicial safeguard, guardianship or curatorship. Patients for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients operated on a reduction nymphoplasty, for uni or bilateral labia minora hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | Change from Baseline 3 yers after surgery
  Questionnaire on the evolution of sexuality. FSFI consists of 19 questions assessing 6 domains: sexual desire, arousal, lubrication, orgasm, sexual satisfaction and pain. It is based on the sexuality of the last 4 weeks. The questions report a score ranging from 0 or 1 to 5 and a different coefficient is assigned to each domain. The sum of these results constitutes the final score, between 2 and 32 with the threshold value defining an alteration of sexuality below 26.5/32.

SECONDARY OUTCOMES:
Body Esteem Scale (BES) | Change from Baseline 3 yers after surgery
  Self-esteem questionnaire BES is composed of 23 questions, rated on a 5-point Likert scale (never, rarely, sometimes, often and always) and divided into 3 items corresponding to different dimensions of self-esteem: appearance, attribution and weight. The score is between 23 and 115, and the higher it is, the higher the body esteem and the appearance evaluated positively

CONTACTS AND LOCATIONS:
Overall Officials: Jenifer SALERNO, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU Nimes, Nîmes, France